CLINICAL TRIAL: NCT04463940
Title: The Origin of Xanthine Oxidase and Its Metabolite, Uric Acid, in Preeclamptic Pregnant Women - A Pilot Study
Brief Title: Xanthine Oxidase and Uric Acid Origin in Preeclamptic Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Simon Shanhav, Dr Simon Shenhav, head of High Risk Pregnancy Unit, Barzilai Medical Center
Other Study IDs: 0024-19-BRZ
Record Dates: First submitted 2020-06-08; First posted 2020-07-09 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Pre-Eclampsia; Hyperuricemia
Keywords: Xanthine oxidase; Uric acid
MeSH Terms: conditions — Pre-Eclampsia; Hyperuricemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Umbilical cord arterial blood: participant's umbilical cord arterial blood will be obtained
  Interventions: Other: No intervention
- Umbilical cord venus blood: participant's umbilical cord Venus blood will be obtained
  Interventions: Other: No intervention
- Maternal blood: participant's blood will be obtained
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Findings regarding the presence of xanthine oxidase and uric acid in different blood locations is important in preeclamptic women. We aim to detecting Xanthine oxidase and uric acid levels in both umbilical cord artery and vein as well as maternal blood (3 "locations") in pregnant women with and without diagnosis of preeclampsia. The study population will be divided into groups matching the three "locations" in order to describe and compare outcome levels.

DETAILED DESCRIPTION:
Significance - findings regarding the presence of xanthine oxidase and uric acid in different blood locations may provide a scientific basis for understanding the source of them in preeclamptic women. Aim - detecting Xanthine oxidase and uric acid levels in both umbilical cord artery and vein as well as maternal blood (3 "locations"). Methods - samples will be collected from pregnant women with and without diagnosis of preeclampsia with blood uric acid > 6 mg/dL. Than the study population will be divided into groups matching the three "locations". The investigators will describe and compare outcome levels (including Xanthine oxidase, uric acid).

ELIGIBILITY:
Inclusion Criteria:

* preeclampsia and none-preeclampsia diagnosed pregnant women.

Exclusion Criteria:

* Known or reported kidney disease.

Ages: 20 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women with and without diagnosis of Pre-Eclampsia and serum Uric Acid greater than 6 mg/dL
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Uric Acid | through study completion, an average of 1 year
  mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Simon Shenhav, Dr, Principal Investigator — Barzilai University Medical Center
Locations (1):
- Barzilai Medical Center, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: Undecided